CLINICAL TRIAL: NCT06792539
Title: A Multi-Center, Prospective, Non-Randomized, Pivotal Trial Evaluating the Safety and Effectiveness of the Polymotion Hip Resurfacing System
Brief Title: Evaluate the Safety and Effectiveness of the Polymotion Hip Resurfacing (PHR) System Compared to Total Hip Arthroplasty
Acronym: PHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JointMedica Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI001
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis of the Hip; Degenerative Joint Disease of Hip; Dysplasia; Hip
Keywords: hip resurfacing; Osteoarthritis of the Hip; deterioration of hip cartilage; Polymotion
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Dislocation | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, non-randomized, propensity score-adjusted, pivotal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Polymotion Hip Resurfacing (PHR) System (Experimental): The investigational device, Polymotion Hip Resurfacing System ("Polymotion" or "PHR"), is a metal-onpolyethylene hip resurfacing device consisting of a metallic femoral component and an acetabular component made of Vitamin E HXLPE with a titanium coating on its bone-contacting surface.
  Both components are designed to be permanently implanted, to achieve reconstructive and functional replacement of the hip joint. The PHR System is intended to offer the traditional benefits of hip resurfacing over total hip arthroplasty, such as bone conservation and restoration of natural biomechanics, without a metal-on-metal articulating surface.
  Interventions: Device: Polymotion Hip Resurfacing (PHR) System

INTERVENTIONS:
Device: Polymotion Hip Resurfacing (PHR) System — Surgical

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of the Polymotion Hip Resurfacing (PHR) System compared to total hip arthroplasty, for adults who require hip resurfacing arthroplasty due to 1) non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, traumatic arthritis, or 2) mild dysplasia/developmental dislocation of the hip (DDH) up to Crowe Grade 1.

DETAILED DESCRIPTION:
The PHR® System is a single-use device consisting of a Cobalt Chromium, bone-cemented femoral head component, and a cementless acetabular component comprising of a Vitamin E polyethylene (Vit E-XPE) bearing with a titanium coating.

The PHR® System is intended for patients who, due to their relatively younger age (under 65) and increased activity level, may not be suitable for traditional total hip arthroplasty due to an increased possibility of requiring future ipsilateral hip joint revision.

Hip Resurfacing Arthroplasty (HRA) is a surgery that has been developed as an alternative to Total Hip Arthroplasty (THA), especially for younger, more active patients. Studies done on past designs of HRA demonstrate the following noteworthy benefits of the HRA procedure when compared with THA: bone conservation, improved gait, higher activity levels, lower rates of dislocations, reduced thigh pain, and reduced alteration in leg length. Hip resurfacing restores the natural shape of the joint meaning better stability, longevity, and higher levels of activity than a traditional hip replacement.

In Total Hip Replacement, the femoral head and neck (ball joint of the hip) is removed and replaced by a long, stemmed device. The procedure is highly successful; however, in some cases the replacement hip joint has the potential to wear out much more quickly in younger, more active patients, leading to revision surgery being required. With the PHR® procedure, your surgeon removes less bone from the femoral head of the femur and retains the femoral neck. The femoral head is shaped to accept a low-wear metal cap. This spherical cap closely matches your anatomy, reducing the risk of dislocation, and offering a broad range of movement and excellent stability. The acetabular socket (cup joint of the hip) is then fitted with a corresponding polyethylene component, significantly reducing potential reactions to metal ions associated with historic Metal-on-Metal hip resurfacing devices.

A comprehensive range of sizes is offered to address the needs of most patients. Both components are designed to be implanted, to achieve reconstructive and functional replacement of the hip joint. The PHR® System is intended to offer the traditional benefits of hip resurfacing over total hip arthroplasties, such as bone conservation and restoration of natural biomechanics, without a metal-on-metal articulating surface.

ELIGIBILITY:
In order to be eligible to participate in this study, subjects must meet all of the following criteria:

1. Requires primary hip resurfacing arthroplasty due to:

   1. non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, traumatic arthritis, or
   2. mild dysplasia/developmental dislocation of the hip (DDH) up to Crowe Grade 1.
2. Harris Hip Score < 70 points.
3. Skeletally mature, age ≥21 and <65 years.
4. Physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.

Subjects who meet any of the following criteria will be excluded from participating in this study:

1. Inadequate bone stock or bone quality to support the device based on a Canal-Bone Ratio (CBR-7) of >0.45.0F
2. Severe osteopenia, a medical history or increased risk of severe osteoporosis or severe osteopenia, a history of fragility fracture, and other conditions that lead to increased bone resorption
3. Osteonecrosis or avascular necrosis (AVN)
4. Multiple cysts of the femoral head (> 1cm) or cysts crossing the head-neck junction
5. Metabolic disorders which may impair bone formation (e.g., osteomalacia, osteogenesis imperfecta, parathyroid disease, rickets, etc.)
6. Severe femoral head deformities that will prevent fixation of the prosthetic resurfacing femoral head
7. Inflammatory arthritis such as rheumatoid arthritis (RA)
8. Severe proximal femoral rotational deformity in whom appropriate combined anteversion of femoral-acetabular construct is unachievable
9. Severe acetabular dysplasia/development dislocation of the hip, defined as Crowe Grade ≥ 2
10. Previous surgical intervention on index hip (e.g., treatment of hip fracture, arthroscopy)
11. Severe medical comorbidities, including:

    1. severe cardiopulmonary disease,
    2. congestive heart failure,
    3. severe liver or kidney dysfunction,
    4. end-stage renal disease,
    5. severe uncontrolled diabetes,
    6. history of IV drug use,
    7. history of hypercoagulable state or pulmonary embolism,
    8. severe lumbar spinal stenosis,
    9. vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or post-operative recovery,
    10. neuropathic arthropathy (Charcot joint),
    11. immunosuppression or other immunodeficiency disorders, e.g., diseases such as Acquired Immune Deficiency Syndrome (AIDS) or post-organ transplant and on high doses of corticosteroids.
12. Incompetent or deficient soft tissue surrounding the joint (e.g., hip abductor muscle deficiency)
13. BMI > 40
14. Active or suspected infection in or around the hip joint
15. Known or suspected metal sensitivity (e.g., jewelry) or allergy to any implant materials
16. Pregnant or plan to become pregnant during the study duration
17. Current smoker

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and clinical effectiveness of the Polymotion Hip Resurfacing System. | 24 months
  The proportion of Polymotion subjects achieving Month-24 composite clinical success (CCS) will be compared to a propensity-score matched total hip arthroplasty control group collected from Rush University Medical Center, with the goal of demonstrating non-inferiority.
  Composite clinical success will be analyzed via Harris Hip Scores measuring pain, activity, and function, absence of device subsidence, progressive radiolucencies, osteolysis or migration through radiographic assessment, and the absence of serious safety events (secondary surgical interventions for the index hip or serious device-related adverse events).

SECONDARY OUTCOMES:
Harris Hip Score, and sub-scores of HHS for pain and function | 24 months
  The Harris Hip Score is used to measure pain severity, function, and absence of deformity.
  Each hip joint is scored on nine parameters, generating a total score representing the severity of the condition. The lower the score the better. The minimum score for each hip is 0 and the maximum is 53, giving a range for the total score of 0 to 106.
SUSHI-University of California Los Angeles (UCLA) Activity Scores | 24 months
  The SUSHI-UCLA Activity Score is a 10-item assessment of physical activity level to assess patients overall state, pain and limitations of their hip.
Hip Disability and Osteoarthritis Outcome Score, Joint Replacement (HOOS JR), and sub-scores of HOOS JR for pain and function | 24 months
  The HOOS JR Survey is a short form of the HOOS that assesses patient pain (2 items), and functions of daily living (4 items).
Forgotten Joint Score | 24 months
  The Forgotten Joint Score consists of 12 questions, scored on a 0-100 scale, intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment.
SF-12 | 24 months
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health.
Radiographic success | 24 months
  Absence of migration, subsidence, and osteyloysis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mont, MD, Principal Investigator — Principal Investigator
Locations (10):
- United States (9):
  - Florida Medical Clinic Orlando Health, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Sinai Hospital / LifeBridge Health, Baltimore, Maryland
  - NYU Longone, New York, New York
  - Joint Implant Surgeons, New Albany, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Midlands Orthopaedics & Neurosurgery, Columbia, South Carolina
  - Hampton Road Orthopaedics, Newport News, Virginia
  - Spokane Joint Replacement Center, Spokane, Washington
- Orthopaedic and Physiotherapy Associates, Paget, Trevelyan, Bermuda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh JA, Schleck C, Harmsen S, Lewallen D. Clinically important improvement thresholds for Harris Hip Score and its ability to predict revision risk after primary total hip arthroplasty. BMC Musculoskelet Disord. 2016 Jun 10;17:256. doi: 10.1186/s12891-016-1106-8. PMID 27286675
- [Background] Treacy RBC, Holland JP, Daniel J, Ziaee H, McMinn DJW. Preliminary report of clinical experience with metal-on-highly-crosslinked-polyethylene hip resurfacing. Bone Joint Res. 2019 Nov 2;8(10):443-450. doi: 10.1302/2046-3758.810.BJR-2019-0060.R1. eCollection 2019 Oct. PMID 31728182
- [Background] Cadossi M, Tedesco G, Sambri A, Mazzotti A, Giannini S. Hip Resurfacing Implants. Orthopedics. 2015 Aug;38(8):504-9. doi: 10.3928/01477447-20150804-07. PMID 26270748
- [Background] Joshi AB, Porter ML, Trail IA, Hunt LP, Murphy JC, Hardinge K. Long-term results of Charnley low-friction arthroplasty in young patients. J Bone Joint Surg Br. 1993 Jul;75(4):616-23. doi: 10.1302/0301-620X.75B4.8331119.
- [Background] Dorr LD, Kane TJ 3rd, Conaty JP. Long-term results of cemented total hip arthroplasty in patients 45 years old or younger. A 16-year follow-up study. J Arthroplasty. 1994 Oct;9(5):453-6. doi: 10.1016/0883-5403(94)90090-6. PMID 7807101
- [Background] Bradley GW, Freeman MA, Revell PA. Resurfacing arthroplasty. Femoral head viability. Clin Orthop Relat Res. 1987 Jul;(220):137-41. PMID 3594982
- [Background] CHARNLEY J. Surgery of the hip-joint: present and future developments. Br Med J. 1960 Mar 19;1(5176):821-6. doi: 10.1136/bmj.1.5176.821. No abstract available. PMID 13809344
- [Background] Hu D, Tie K, Yang X, Tan Y, Alaidaros M, Chen L. Comparison of ceramic-on-ceramic to metal-on-polyethylene bearing surfaces in total hip arthroplasty: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2015 Feb 3;10:22. doi: 10.1186/s13018-015-0163-2. PMID 25645809
- [Background] Varnum C. Outcomes of different bearings in total hip arthroplasty - implant survival, revision causes, and patient-reported outcome. Dan Med J. 2017 Mar;64(3):B5350. PMID 28260601
- [Background] Campbell P, Ebramzadeh E, Nelson S, Takamura K, De Smet K, Amstutz HC. Histological features of pseudotumor-like tissues from metal-on-metal hips. Clin Orthop Relat Res. 2010 Sep;468(9):2321-7. doi: 10.1007/s11999-010-1372-y. PMID 20458645
- [Background] Corradi M, Daniel J, Ziaee H, Alinovi R, Mutti A, McMinn DJ. Early markers of nephrotoxicity in patients with metal-on-metal hip arthroplasty. Clin Orthop Relat Res. 2011 Jun;469(6):1651-9. doi: 10.1007/s11999-010-1682-0. PMID 21108029
- [Background] Visuri T, Borg H, Pulkkinen P, Paavolainen P, Pukkala E. A retrospective comparative study of mortality and causes of death among patients with metal-on-metal and metal-on-polyethylene total hip prostheses in primary osteoarthritis after a long-term follow-up. BMC Musculoskelet Disord. 2010 Apr 23;11:78. doi: 10.1186/1471-2474-11-78. PMID 20416065
- [Background] Smith AJ, Dieppe P, Porter M, Blom AW; National Joint Registry of England and Wales. Risk of cancer in first seven years after metal-on-metal hip replacement compared with other bearings and general population: linkage study between the National Joint Registry of England and Wales and hospital episode statistics. BMJ. 2012 Apr 3;344:e2383. doi: 10.1136/bmj.e2383. PMID 22490979
- [Background] Kendal AR, Prieto-Alhambra D, Arden NK, Carr A, Judge A. Mortality rates at 10 years after metal-on-metal hip resurfacing compared with total hip replacement in England: retrospective cohort analysis of hospital episode statistics. BMJ. 2013 Nov 27;347:f6549. doi: 10.1136/bmj.f6549. PMID 24284336
- [Background] Gill HS, Grammatopoulos G, Adshead S, Tsialogiannis E, Tsiridis E. Molecular and immune toxicity of CoCr nanoparticles in MoM hip arthroplasty. Trends Mol Med. 2012 Mar;18(3):145-55. doi: 10.1016/j.molmed.2011.12.002. Epub 2012 Jan 12. PMID 22245020
- [Background] Catalani S, Rizzetti MC, Padovani A, Apostoli P. Neurotoxicity of cobalt. Hum Exp Toxicol. 2012 May;31(5):421-37. doi: 10.1177/0960327111414280. Epub 2011 Jul 5. PMID 21729976
- [Background] Gessner BD, Steck T, Woelber E, Tower SS. A Systematic Review of Systemic Cobaltism After Wear or Corrosion of Chrome-Cobalt Hip Implants. J Patient Saf. 2019 Jun;15(2):97-104. doi: 10.1097/PTS.0000000000000220. PMID 26076080
- [Background] McMinn D, Daniel J. History and modern concepts in surface replacement. Proc Inst Mech Eng H. 2006 Feb;220(2):239-51. doi: 10.1243/095441105X68944. PMID 16669391
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Pivec R, Johnson AJ, Mears SC, Mont MA. Hip arthroplasty. Lancet. 2012 Nov 17;380(9855):1768-77. doi: 10.1016/S0140-6736(12)60607-2. Epub 2012 Sep 26. PMID 23021846
- [Background] Okike K, King RK, Merchant JC, Toney EA, Lee GY, Yoon HC. Rapidly Destructive Hip Disease Following Intra-Articular Corticosteroid Injection of the Hip. J Bone Joint Surg Am. 2021 Nov 17;103(22):2070-2079. doi: 10.2106/JBJS.20.02155. PMID 34550909
- [Background] Stevenson DA, Mineau G, Kerber RA, Viskochil DH, Schaefer C, Roach JW. Familial predisposition to developmental dysplasia of the hip. J Pediatr Orthop. 2009 Jul-Aug;29(5):463-6. doi: 10.1097/BPO.0b013e3181aa586b. PMID 19568018
- [Background] Hoaglund FT, Healey JH. Osteoarthrosis and congenital dysplasia of the hip in family members of children who have congenital dysplasia of the hip. J Bone Joint Surg Am. 1990 Dec;72(10):1510-8. PMID 2254359
- [Background] Shaw BA, Segal LS; SECTION ON ORTHOPAEDICS. Evaluation and Referral for Developmental Dysplasia of the Hip in Infants. Pediatrics. 2016 Dec;138(6):e20163107. doi: 10.1542/peds.2016-3107. Epub 2016 Nov 21. PMID 27940740
- [Background] Hoaglund FT, Kalamchi A, Poon R, Chow SP, Yau AC. Congenital hip dislocation and dysplasia in Southern Chinese. Int Orthop. 1981;4(4):243-6. doi: 10.1007/BF00266064. PMID 7228460
- [Background] Skirving AP, Scadden WJ. The African neonatal hip and its immunity from congenital dislocation. J Bone Joint Surg Br. 1979 Aug;61-B(3):339-41. doi: 10.1302/0301-620X.61B3.479257.
- [Background] Coleman SS. Congenital dysplasia of the hip in the Navajo infant. Clin Orthop Relat Res. 1968 Jan-Feb;56:179-93. No abstract available. PMID 5652776
- [Background] Reidy M, Collins C, MacLean JGB, Campbell D. Examining the effectiveness of examination at 6-8 weeks for developmental dysplasia: testing the safety net. Arch Dis Child. 2019 Oct;104(10):953-955. doi: 10.1136/archdischild-2018-316520. Epub 2018 Dec 5. PMID 30518519
- [Background] Lehmann HP, Hinton R, Morello P, Santoli J. Developmental dysplasia of the hip practice guideline: technical report. Committee on Quality Improvement, and Subcommittee on Developmental Dysplasia of the Hip. Pediatrics. 2000 Apr;105(4):E57. doi: 10.1542/peds.105.4.e57. PMID 10742378
- [Background] Bialik V, Bialik GM, Blazer S, Sujov P, Wiener F, Berant M. Developmental dysplasia of the hip: a new approach to incidence. Pediatrics. 1999 Jan;103(1):93-9. doi: 10.1542/peds.103.1.93. PMID 9917445
- [Background] Dunn PM. The anatomy and pathology of congenital dislocation of the hip. Clin Orthop Relat Res. 1976 Sep;(119):23-7. PMID 954316
- [Background] Cohen-Rosenblum A, Cui Q. Osteonecrosis of the Femoral Head. Orthop Clin North Am. 2019 Apr;50(2):139-149. doi: 10.1016/j.ocl.2018.10.001. Epub 2019 Feb 12. PMID 30850073
- [Background] Guerado E, Caso E. The physiopathology of avascular necrosis of the femoral head: an update. Injury. 2016 Dec;47 Suppl 6:S16-S26. doi: 10.1016/S0020-1383(16)30835-X. PMID 28040082
- [Background] Eriksson JK, Neovius M, Ernestam S, Lindblad S, Simard JF, Askling J. Incidence of rheumatoid arthritis in Sweden: a nationwide population-based assessment of incidence, its determinants, and treatment penetration. Arthritis Care Res (Hoboken). 2013 Jun;65(6):870-8. doi: 10.1002/acr.21900. PMID 23281173
- [Background] Di Giuseppe D, Alfredsson L, Bottai M, Askling J, Wolk A. Long term alcohol intake and risk of rheumatoid arthritis in women: a population based cohort study. BMJ. 2012 Jul 10;345:e4230. doi: 10.1136/bmj.e4230. PMID 22782847
- [Background] Hunter TM, Boytsov NN, Zhang X, Schroeder K, Michaud K, Araujo AB. Prevalence of rheumatoid arthritis in the United States adult population in healthcare claims databases, 2004-2014. Rheumatol Int. 2017 Sep;37(9):1551-1557. doi: 10.1007/s00296-017-3726-1. Epub 2017 Apr 28. PMID 28455559
- [Background] Myasoedova E, Crowson CS, Kremers HM, Therneau TM, Gabriel SE. Is the incidence of rheumatoid arthritis rising?: results from Olmsted County, Minnesota, 1955-2007. Arthritis Rheum. 2010 Jun;62(6):1576-82. doi: 10.1002/art.27425. PMID 20191579
- [Background] Bohler C, Weimann P, Alasti F, Smolen JS, Windhager R, Aletaha D. Rheumatoid arthritis disease activity and the risk of aseptic arthroplasty loosening. Semin Arthritis Rheum. 2020 Apr;50(2):245-251. doi: 10.1016/j.semarthrit.2019.07.011. Epub 2019 Aug 1. PMID 31471012
- [Background] Swarup I, Sutherland R, Burket JC, Figgie MP. Total hip arthroplasty in young patients with post-traumatic arthritis of the hip. Hip Int. 2017 Nov 21;27(6):546-550. doi: 10.5301/hipint.5000499. Epub 2017 May 23. PMID 28574124
- [Background] Long H, Liu Q, Yin H, Wang K, Diao N, Zhang Y, Lin J, Guo A. Prevalence Trends of Site-Specific Osteoarthritis From 1990 to 2019: Findings From the Global Burden of Disease Study 2019. Arthritis Rheumatol. 2022 Jul;74(7):1172-1183. doi: 10.1002/art.42089. Epub 2022 Jun 2. PMID 35233975
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- See also: Osteoarthritis. — http://dx.doi.org/10.21037/aoj.2019.12.08
- See also: Related Info — https://www.mayoclinic.org/diseases-conditions/osteoarthritis/symptoms-causes/syc-20351925